CLINICAL TRIAL: NCT02889536
Title: Living With a Parastomal Bulge - a Phenomenological-hermeneutic Study of Patients Lived Experiences
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Marianne Krogsgaard, RN, MHS, Rigshospitalet, Denmark
Other Study IDs: PreParE-qualitative
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Ostomy; Hernia; Signs and Symptoms
Keywords: parastomal hernia; ostomy; qualitative; phenomenological-hermeneutic research; symptoms; parastomal bulging
MeSH Terms: conditions — Hernia; Signs and Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Focus group interview, stoma clinics: Qualitative data collection. Patients attending stoma clinics in the capital region
  Interventions: Other: Focus group interviews
- Focus group interview, referred: Qualitative data collection. Patients referred to repair surgery at a specific hospital in the capital region
  Interventions: Other: Focus group interviews

INTERVENTIONS:
Other: Focus group interviews — Focus group interviews. Two groups with patients referred to repair of parastomal bulging and three groups with patients attending the outpatient stoma clinics
  Other Names: Qualitative data collection

SUMMARY:
A parastomal bulge (PB) is a frequent long-term complication after stoma formation. Most parastomal bulging occurs within two years of stoma formation but is seen up to 20 years post-surgery. A bulge may be relatively obvious or extremely difficult to diagnose, and descriptions of symptoms vary from 'asymptomatic', 'symptomatic' to 'high symptom load'. Previous studies report that quality of life as well as physical, psychological and social function are affected in patients with parastomal bulging. However, there is a lack of knowledge of patients' lived experiences with parastomal bulging. Insight into patients' experiences of symptoms in relation to parastomal bulging and the impact on everyday life may help identify issues of importance from the patient perspective. This, in turn, may help professionals to better understand and support patients with PB, and be of help when identifying patients' symptoms and determining relevant treatment strategies.

DETAILED DESCRIPTION:
Stoma formation is a commonly performed procedure in colorectal surgery as part of treatment for malignant- and inflammatory bowel disease. A parastomal bulge (PB) is a frequent long-term complication with an incidence varying from 4% to more than 40% depending on ostomy type, follow-up and definitions.

A bulge may be relatively obvious or extremely difficult to diagnose. Most parastomal bulging occurs within two years of stoma formation but is seen up to 20 years post-surgery. Despite advances in primary surgical and repair techniques a rising incidence of parastomal bulging is expected in the future due to increased survival of cancer patients with an ostomy and limited dissemination of new techniques. Approximately one in three patients with a parastomal hernia requires a surgical hernia repair. However, the majority of patients are referred to non-surgical treatment by the enterostomal therapist in the outpatient clinic or do not seek professional help to manage the bulge. Previous studies report that quality of life as well as physical, psychological and social function are affected in patients with parastomal bulging.

Descriptions of symptoms vary from 'asymptomatic', 'symptomatic' to 'high symptom load'. Most frequently reported symptoms include ostomy leakage, skin problems, difficulty with ostomy appliance, limitation of activity, difficulty with clothing, cosmetic complaints, social restriction, erratic action of the stoma and a bearing down sensation at the site of the stoma. Rare, but serious complications include complete obstruction, strangulation or incarceration. However, there is a lack of knowledge of patients' lived experiences with parastomal bulging. Insight into patients' experiences of symptoms in relation to parastomal bulging and the impact on everyday life may help identify issues of importance from the patient perspective. This, in turn, may help professionals to better understand and support patients with PB, and be of help when identifying patients' symptoms and determining relevant treatment strategies.

Purpose: The aim is to study stoma patients experiences of parastomal bulging and symptoms in everyday life (in relation to an ileostomy and colostomy)

ELIGIBILITY:
Inclusion Criteria:

Permanent or temporary active sigmoidostomy, transversostomy, jejunostomy or ileostomy

PB diagnosed by stoma care nurse

Ability to speak and understand Danish

Exclusion Criteria:

Previous surgical repair for PB

Major incisional abdominal hernias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stoma patients that are routinely followed for at least one year post surgery by stoma care nurses (SCNs) at the outpatient stoma clinics at the five hospitals within the region.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Patients' experiences of symptoms in relation to parastomal bulging and the impact on everyday life | 1 day
  A funnel-based interview approach will be used, allowing for a less structured, open beginning moving to a more structured ending ensuring that the research question will be answered

CONTACTS AND LOCATIONS:
Overall Officials: Thordis Thomsen, PhD, RN, Study Chair — Abdominal Centre, Rigshospitalet, Copenhagen Denmark
Locations (1):
- Marianne Krogsgaard, Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No